CLINICAL TRIAL: NCT03174821
Title: The Impact of Insulin Pump Therapy to Oxidative Stress in Patients With Diabetic Nephropathy
Brief Title: Effect Insulin Pump Therapy to Patients With Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng Lv, Principal investigator, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPT-OX-10
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Insulin Pump Therapy in Treating Diabetic Nephropathy
Keywords: Diabetic nephropathy; Insulin pump intensive therapy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Insulin Infusion Systems

STUDY DESIGN:
Intervention Model Description: Normal group (NC) and Type 2 diabetic (DM) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin pump therapy (Experimental): The total requisite amount=0.44×weight (Kg); The preprandial and basal amount respectively took up 50% of integral dose.15 minutes before meal the preprandial insulin was equally given by 3 times. The basal insulin was pumped at 00:00-3:00，3:00-8:00，8:00-14:00，14:00-20:00，20:00-24:00.
  Interventions: Device: Insulin pump
- Normal control (No Intervention): The subjects were asked to maintain normal diet and lifestyle until the end of the observation period.

INTERVENTIONS:
Device: Insulin pump — Blood glucose management device
  Other Names: Diabetes insulin pump
  Arms: Insulin pump therapy

SUMMARY:
The recent study suggested that oxidative stress resulting from increased production of reactive oxygen species (ROS) plays a crucial role in the development of diabetic complications. The researches aim to monitor the level of oxidative stress of patient in different stage of diabetic nephropathy before and after insulin pump therapy.

DETAILED DESCRIPTION:
Worldwidely, about 30% of Type 1 Diabetes Mellitus (T1DM) and 20%-50% of T2DM patients suffered diabetic nephropathy (DN). Oxidative stress resulting from increased production of reactive oxygen species (ROS) plays a crucial role in the development of diabetic complications. Insulin pump therapy is better than subcutaneous injection in terms of the drug safety and effectiveness. The researches aim to monitor the level of oxidative stress of patient in different stage of diabetic nephropathy before and after insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

Diabetic patients with fasting plasma glucose (FPG) ≥10mmol/l and/or 2 hours' plasma glucose (2hPG) ≥15mmol/l.

Exclusion Criteria:

Diabetic patients who

1. using antioxidant drugs within one month;
2. accompanied with acute and chronic severe complications, fever, malignant tumor, nephritis, congestive heart failure.
3. accompanied with diabetic ketosis, ketoacidosis, severe hypoglycemia, hyperosmolar hyperglycemic state;
4. with other endocrine diseases, autoimmune diseases, or connective tissue diseases;
5. having history of infection within 1 month;
6. having drug or alcohol dependence;
7. severe hypoxia and stress state (e.g., cardiovascular events, trauma, surgery, and consumptive disease, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-10-20 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2014-05-16 (Actual)

PRIMARY OUTCOMES:
The change of 8-hydroxy-deoxyguanosine (8-OHdG) | 2 weeks
  The change of 8-hydroxy-deoxyguanosine (8-OHdG) in serum of diabetic patients with diabetic nephropathy (DN)

SECONDARY OUTCOMES:
The change of 3-nitrotyrosine (3-NT) | 2 weeks
  The change of 3-nitrotyrosine (3-NT) in serum
The change of glutathione (GSH) | 2 weeks
  The change of glutathione (GSH) in serum
The change of superoxide dismutase (SOD) | 2 weeks
  The change of superoxide dismutase (SOD) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Min Liu, Study Chair — Center for Drug Evaluation, China food and Drug Administration

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) was not allowed to use outside this research.

REFERENCES:
- [Derived] Zhang XG, Zhang YQ, Cheng QP, Cao Y, Sun JM, Lv XF. The impact of insulin pump therapy to oxidative stress in patients with diabetic nephropathy. Eur J Med Res. 2018 Feb 12;23(1):7. doi: 10.1186/s40001-018-0304-2. PMID 29433562